CLINICAL TRIAL: NCT02523742
Title: Study of the Hemispheric Specialization for Language in Subjects With Neuropsychiatric Disorders Compared to Control Subjects
Acronym: BIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 05-097
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2015-08

CONDITIONS: Neuropsychiatric Disorders
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuropsychiatric Disorders (Other): Neuropsychiatric Disorders patients
  Interventions: Device: IMRf; Other: language task and a reference task (rest and Tamil)
- Healthy volunteers (Other): control subjects matched to patients by age, sex, socio-cultural level and laterality
  Interventions: Device: IMRf; Other: language task and a reference task (rest and Tamil)

INTERVENTIONS:
Device: IMRf
Other: language task and a reference task (rest and Tamil)

SUMMARY:
Recently, we have shown functional resonance imaging (fMRI) that variations in signal induced by a language task were significantly lower in a semantic region of the left hemisphere (comprised of that part pars triangularis of the inferior frontal gyrus and the temporal gyri medium and angular) in schizophrenic patients compared with controls matched for age, sex, level of education and handedness.

Investigators wish to test the hypothesis that functional modification of the hemispherical specialization is specific language and also specific for schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* patients under 65 years
* Schizophrenics, bipolar or schizoaffective (DSM IV)
* Patients who signed informed consent

Exclusion Criteria:

* Women with childbearing potential without effective contraception or positive pregnancy test.
* Contra-indications to fMRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2013-11-19 (Actual); Study Completion 2015-04-23 (Actual)

PRIMARY OUTCOMES:
variation in signal (SPM99) during a language task compared to a reference task (rest or Tamil) in fMRI in anatomical regions of interest | baseline